CLINICAL TRIAL: NCT06520527
Title: Comparison of the Effectiveness of Sambiloto Herbs (Andrographis Paniculata) and Brisk Walking Exercise on Blood Pressure of Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Palangka Raya (Other)
Responsible Party: Principal Investigator, Agnes Veronica Agustin, Agnes Veronica Agustin, Universitas Palangka Raya
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2504031945
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: MeSH
Keywords: Obese
MeSH Terms: conditions — Obesity | interventions — Andrographis paniculata extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Brisk Walking Exercise (Experimental): Moderate activity that uses brisk walking techniques for 30 minutes at an average speed of up to 5 km/h or 100 steps per minute.a
  Interventions: Behavioral: Brisk Walking Exercise
- Andrographis Paniculata (Experimental): Jamu Sambiloto is herbal medicine obtained through products that already have a distribution permit and have a distribution permit registration number, with a consumption dose of 1 capul / day or 350 grams for 7 consecutive days.
  Interventions: Dietary Supplement: Andrographis paniculata
- Combination (Experimental): Moderate activity that uses brisk walking techniques for 30 minutes at an average speed of up to 5 km/h or 100 steps per minute.a
  Jamu Sambiloto is herbal medicine obtained through products that already have a distribution permit and have a distribution permit registration number, with a consumption dose of 1 capul / day or 350 grams for 7 consecutive days.
  Interventions: Other: Combination
- Control (No Intervention): Obese with no intervention
- Normal (No Intervention): Normal with no intervention

INTERVENTIONS:
Dietary Supplement: Andrographis paniculata — Jamu Sambiloto is herbal medicine obtained through products that already have a distribution permit and have a distribution permit registration number, with a consumption dose of 1 capul / day or 350 grams for 7 consecutive days.
  Arms: Andrographis Paniculata
Behavioral: Brisk Walking Exercise — Moderate activity that uses brisk walking techniques for 30 minutes at an average speed of up to 5 km/h or 100 steps per minute.
  Arms: Brisk Walking Exercise
Other: Combination — Moderate activity that uses brisk walking techniques for 30 minutes at an average speed of up to 5 km/h or 100 steps per minute.
  Jamu Sambiloto is herbal medicine obtained through products that already have a distribution permit and have a distribution permit registration number, with a consumption dose of 1 capul / day or 350 grams for 7 consecutive days.
  Arms: Combination

SUMMARY:
Problem Formulation

1. Is there an effect of giving jamu sambiloto (Andrographis paniculata) on blood pressure in obese people in Jekan Raya District?
2. Is there an effect of brisk walking exercise on blood pressure in obese people in Jekan Raya District?
3. Is there an effect of brisk walking exercise and combined administration of jamu sambiloto (Andrographis paniculata) on blood pressure in obese people in Jekan Raya District?
4. Is there a difference in effectiveness between the administration of jamu sambiloto (Andrographis paniculata) and brisk walking exercise and the combination on blood pressure in obese people in Jekan Raya District?

Research Objectives

General Objective:

This study aims to determine the difference in effectiveness between the administration of jamu sambiloto (Andrographis paniculata) and brisk walking exercise on blood pressure in obese people in Jekan Raya District.

Specific Objectives:

This study specifically aims to:

1. Knowing the effect on blood pressure of obese people in Jekan Raya District before and after giving Jamu Sambiloto (Andrographis paniculata).
2. Knowing the effect on blood pressure of obese people in Jekan Raya District before and after doing Brisk Walking Exercise.
3. Knowing the effect before and after giving Jamu Sambiloto (Andrographis paniculata) and Brisk Walking Exercise on Blood Pressure in obese people in Jekan Raya District.

DETAILED DESCRIPTION:
This type of research uses the Quasi Experimental method type Non-equivalent control group design, with a research design in the form of two group pre test and post test design, in this study there are two groups that will be measured pretest before intervention and post test after intervention and 1 control group without being given intervention. The intervention group is divided into two groups, namely the group given the sambiloto herbal medicine, and the group given the Brisk Walking Exercise treatment. Quasi-experimental research design with research design in the form of two group pre test and post test design.

ELIGIBILITY:
Inclusion criteria in this study are:

Body Mass Index (BMI) ≥ 25 kg/m2 (Obesity 1) Blood pressure does not exceed 139/89 mmHg (High Normal) Adult age (19-39 years) Willing to be a respondent with informed consent Have health insurance coverage

Exclusion Criteria

Exclusion criteria in this study are:

Not in place or out of town during the study Experiencing illness that cannot carry out research interventions and data collection Resign during the study Routine exercise (Exercise every day less than 6000 steps). Taking anti-hypertensive drugs regularly Pregnant and breastfeeding mothers Routinely consume jamu sambiloto History of bone and joint disease that prevents physical activity History of cardiovascular or kidney disease

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-21 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Systole and Diastole Differences | 7 consecutive days
  Difference in Systole and Diastole before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sports Facilities, Palangkaraya, Central Kalimantan, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided